CLINICAL TRIAL: NCT05210244
Title: Acute Effects of Beetroot Juice Supplementation Among Neuromuscular Performance in Amateur Climbers
Brief Title: Acute Beetroot Juice Supplementation in Amateur Climbers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Francisco de Vitoria (Other)
Responsible Party: Principal Investigator, Luis Berlanga, Principal Investigator, Universidad Francisco de Vitoria
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UFV2020-44
Record Dates: First submitted 2022-01-25; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Dietary Supplement; Sport Performance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BJ supplementation (Experimental)
  Interventions: Dietary Supplement: Beetroot Juice (BJ) acute supplementation
- PLA supplementation (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo Juice (PLA) acute supplementation

INTERVENTIONS:
Dietary Supplement: Beetroot Juice (BJ) acute supplementation — One serving of 70 mL of BJ (6.4 mmol of NO3) 3h before initiating the testing session
  Arms: BJ supplementation
Dietary Supplement: Placebo Juice (PLA) acute supplementation — One serving of 70 mL of juice (0.005 mmol of NO3) 3h before initiating the testing session
  Arms: PLA supplementation

SUMMARY:
Whereas beetroot juice (BJ) supplementation is shown to increase physical performance in endurance activities, its benefits in neuromuscular function and strength performance has been barely studied. In this cross-over randomized placebo-controlled study, we investigated the effects of BJ acute supplementation in improving neuromuscular performance in amateur climbers

ELIGIBILITY:
Inclusion Criteria:

* more than 18 years
* active climbing for, at least, last 6 months

Exclusion Criteria:

* smoking
* contraindications to BJ diet
* physical limitations, health problems, or musculoskeletal injuries

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Changes in rate of force development (N/s) at 50, 100 and 200 ms; and at 95% of maximal force | 1 week
  Using a force sensor

SECONDARY OUTCOMES:
Changes in nitrites and nitrates levels in saliva (μmol/L) | 1 week
  Using specific kit ELISA analysis
Changes in maximal number of pull-ups | 1 week
Changes in maximal isometric handgrip strength (kg) | 1 week
  Using a dynamometer
Changes in maximal jump height (cm) | 1 week
  Maximal jump height using a contact platform

CONTACTS AND LOCATIONS:
Overall Officials: Luis Berlanga, Principal Investigator — Universidad Francisco de Vitoria
Locations (1):
- Universidad Francisco de Vitoria, Pozuelo de Alarcón, Madrid, Spain